CLINICAL TRIAL: NCT06415292
Title: A Clinical Study to Assess the Barrier Impact of Winlevi
Brief Title: A Study to Evaluate the Impact of Clascoterone 1% Cream on Skin Barrier Properties in Acne Prone Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: DCS-94-23
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Clascoterone

STUDY DESIGN:
Intervention Model Description: Patients were randomized to apply treatment (winlevi 1%) to one side of the face and the other side of the face remained untreated
Who Masked: Investigator, Outcomes Assessor
Masking Description: The Outcomes Assessor/Investigator was blinded to which side of the face received the treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Winlevi (clascoterone) 1% treated (Experimental): Splitface design- Subjects applied Winlevi (clascoterone) cream 1%, twice daily to the randomized half face following cleansing, every morning and evening.
  Interventions: Drug: Winlevi (clascoterone) 1% cream
- Splitface design- No study product (No Intervention): Splitface design-no study product was applied to the untreated side of the face

INTERVENTIONS:
Drug: Winlevi (clascoterone) 1% cream — Splitface design- Subjects applied Winlevi (clascoterone) cream 1%, twice daily to the randomized half face following cleansing, every morning and evening.
  Arms: Winlevi (clascoterone) 1% treated

SUMMARY:
Acne medications are a common source of facial dryness resulting in skin barrier damage and poor patient compliance. Retinoids and benzoyl peroxide are some of the most frequently prescribed and effective acne medications, however, dryness is an unwanted side effect. A new acne medication, 1% clascoterone, has been placed in a novel vehicle for excellent drug delivery in combination with excellent barrier properties. The barrier properties of 1% clascoterone have never been demonstrated. This study is aimed at better understanding the positive barrier effects of 1% clascoterone.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who self identify as having sensitive acne prone skin.
2. Female or male subjects 18+ years of age.
3. Subjects with Fitzpatrick skin types I-VI.
4. Subject agrees not to introduce any new colored cosmetics (lipsticks, eye shadows, facial foundations, blush, powder) or skin care products during the study.
5. Subjects must be willing to use only a cleanser and sunscreen on the entire face and no other skin care products.
6. Subjects must be willing to use the Winlevi study product to designated half face. No other topical acne treatment products on the entire face for the 2 week duration of the study.
7. Subject has signed an Informed Consent Form in compliance with 21CFR Part 50: "Protection of Human Subjects."
8. Subject is dependable and able to follow directions and is willing to comply with the schedule of visits.
9. Subject is in generally good physical and mental health.

Exclusion Criteria:

1. Any dermatological disorder, which in the investigator's opinion, may interfere with the accurate evaluation of the subject's skin characteristics, except for the conditions associated with sensitive skin.
2. Subjects who are not willing to use only the assigned study product and nothing else one randomized half face, except for cleanser and sunscreen that must remain unchanged during the study. Moisturizers or topical acne treatment products should not be used during the 2 week study period on either side of the face.
3. Subjects who do not agree to refrain from direct sun exposure during the study duration.
4. Subjects who have demonstrated a previous hypersensitivity reaction to any of the ingredients of the study products.
5. Subjects, who are pregnant, breast feeding, or planning a pregnancy.
6. Subjects with clinically significant unstable medical disorders.
7. Subjects who are unwilling or unable to comply with the requirements of the protocol.
8. Subjects who have history of a psychological illness or condition that would interfere with their ability to understand and follow the requirements of the study.
9. Subjects who are currently participating in any other clinical study.
10. Subjects with any planned surgeries and/or invasive medical procedures during the course of the study.
11. Subjects who currently or frequently use high doses of anti-inflammatory drugs for a defined medication condition. Aspirin use should not exceed 2 tablets (650 mg) per day.
12. Subjects currently receiving any anticancer, immunosuppressive treatments/ medications (e.g., azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara.), or radiation as determined by the initial paperwork.
13. Subjects with a history of immunosuppression/immune deficiency disorders (including (HIV infection or AIDS) or currently using immunosuppressive medications (e.g., azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara) and/or radiation as determined by study documentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2023-12-16 (Actual); Study Completion 2023-12-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Consulting Services, PLLC, High Point, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Split face
Groups:
- Winlevi (Clascoterone) 1% Treated: This study involved 50 subjects. Splitface design- Subjects applied Winlevi(clascoterone) cream 1%, twice daily to the randomized half face following cleansing, everymorning and evening. No study product was applied to the untreated side of the face
Period: Overall Study
Arm/Group | Winlevi (Clascoterone) 1% Treated
Started | 50; 100 Split face
Winlevi (Clascoterone) 1% Un-treated Side (UT) | 50; 50 Split face
Winlevi (Clascoterone) 1% Treated Side (T) | 50; 50 Split face
Completed | 49; 98 Split face
Not Completed | 1; 2 Split face

BASELINE CHARACTERISTICS:
Groups:
- Winlevi (Clascoterone) 1% Treated: Winlevi (clascoterone) 1% cream: Split face. Blinded study treatment product to be applied to the randomized half face
Arm/Group | Winlevi (Clascoterone) 1% Treated
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 1
  African Americans | 19
  Caucasians | 30

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint is the Change in Corneometry Reading Between the Two Sides of the Face Treated With Winlevi Versus no Treatment.
Description: The Corneometer measures skin hydration with a range of 0- 1000 MicroSiemens, where 0 is lowest and 1000 is highest hydration
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: microSiemens (μS)
Groups:
- Winlevi (Clascoterone) 1% Un-treated Side (UT): Splitface design-no study product was applied to the untreated side of the face
- Winlevi (Clascoterone) 1% Treated Side (T): Splitface design- Subjects applied Winlevi (clascoterone) cream 1%, twice daily to the randomized half face following cleansing, every morning and evening.
Arm/Group | Winlevi (Clascoterone) 1% Un-treated Side (UT) | Winlevi (Clascoterone) 1% Treated Side (T)
Number analyzed (Participants) | 50 | 50
microSiemens (μS) | 131.27 (42.92) | 113.94 (36.61)
Statistical Analysis 1: Comparison: Winlevi (Clascoterone) 1% Un-treated Side (UT); Test type: Superiority; p < 0.001, t-test, 2 sided — The P-value reported here is the calculated p-value. The p-value theshold for significance was p =0.05

2. Secondary Outcome: Change in TEWL Reading Between the Two Sides of the Face Treated With Winlevi Versus no Treatment
Description: The instrument measures trans epidermal water loss (abbreviated as TEWL) which ranges from minimum 0 (no trans epidermal water loss) to maximum 100 (high trans epidermal water loss)
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: g/h/m²
Groups:
- Winlevi Un-treated Side (UT): Splitface design-no study product was applied to the untreated side of the face
- Winlevi Treated Side (T): Splitface design- Subjects applied Winlevi (clascoterone) cream 1%, twice daily to the randomized half face following cleansing, every morning and evening.
Arm/Group | Winlevi Un-treated Side (UT) | Winlevi Treated Side (T)
Number analyzed (Participants) | 50 | 50
g/h/m² | 9.94 (2.59) | 9.92 (2.88)

ADVERSE EVENTS:
Time Frame: 2 Weeks
Description: There was only one patient that report Covid 19 during the study, this patient applied winlevi to one side of the face and the other side was left untreated.
Arm/Group | Winlevi (Clascoterone) 1% Treated
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 1/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Winlevi (Clascoterone) 1% Treated (N=50)
Covid 19 (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT06415292/Prot_SAP_000.pdf